CLINICAL TRIAL: NCT02249975
Title: Efficacy of CryoBalloon Focal Ablation System on Human Esophageal Barrett's Epithelium
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pentax Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP-0004.A
Record Dates: First submitted 2014-09-24; First posted 2014-09-26 (Estimated); Last update posted 2022-04-28 (Actual); Status verified 2018-02

CONDITIONS: Barrett's Esophagus
MeSH Terms: conditions — Barrett Esophagus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- C2 CryoBalloon Focal Ablation System (Experimental): Cryoballoon ablation will be performed on patients with Barrett's Esophagus.
  Interventions: Device: C2 CryoBalloon Focal Ablation System

INTERVENTIONS:
Device: C2 CryoBalloon Focal Ablation System — The C2 Focal Cryoablation Device will be used for the treatment of islands of BE in real patient care. Ablation at 10 seconds will be tested and post-ablation symptoms related to the Cryoballoon Focal Ablation will be recorded. At 12 weeks, the patient will receive a follow-up endoscopy and biopsy samples will be taken.
  Biopsy samples will be evaluated for the presence of residual Barrett's Esophagus. Through evaluation of the histological results, treatment parameters for the ablation of human esophageal epithelium will be better understood.
  Evaluations include, but are not limited to the following:
  * Device malfunctions
  * Adverse events
  * Patient Pain
  * Histological evaluation of treatment zone at 12 weeks for presence of residual Barrett's Esophagus.

SUMMARY:
The purpose of this study is to assess the efficacy and performance of the C2 Focal Cryoablation System in patients with BE.

DETAILED DESCRIPTION:
The purpose of this study is to assess the efficacy and performance of the C2 Focal Cryoablation System in patients with BE. The study will involve up to 50 subjects with each subject receiving cryoablation therapy of all visible BE using the C2 System Focal Ablation System. Length of ablation will be 10 seconds. The ablations will be performed on Barrett's epithelium with a maximal length of 6 cm.

At the time of endoscopic follow up, biopsies of the treated area will be taken and submitted for analysis according to Histopathology Protocol.

This study is:

* Prospective
* Multi-center
* Non-randomized

ELIGIBILITY:
Criteria Inclusion Criteria

* Patients with known Barrett's esophagus, with an indication for ablation therapy during which the cryoablation may be performed.
* Patient is 18 to 80 years of age at the time of consent (inclusive).
* Patient has provided written Informed Consent (IC) using an Informed Consent Form (ICF) that has been approved by the Institution's reviewing IRB/EC.
* Patient is willing and able to comply with all Clinical Investigation Plan (CIP) requirements.
* Patient is deemed operable per standard institutional criteria.
* BE lesion length <6cm excluding visible BE islands, and Prague Classification C ≥ 0 / M ≥ 0.
* One of the following: Flat LGD, Flat HGD, Residual BE after EMR for visible lesions (containing any degree of dysplasia or low-risk early adenocarcinoma (i.e.: not poorly differentiated, negative vertical (deep) resection margins, absence of (lympho)vascular invasion), Residual BE after a single circumferential RFA (performed for indications listed above: i-iii)
* BE lesion within the treatment zone should be flat

Exclusion Criteria

* Esophageal stenosis preventing advancement of a therapeutic endoscope within 4 cm of treatment zone.
* Patient has a known history of unresolved drug or alcohol dependency that would limit ability to comprehend or follow instructions related to informed consent, post treatment instructions or follow-up guidelines.
* Patient refuses or is unable to provide written informed consent.
* Patients that are pregnant.
* Patient with endoscopically active inflammation in the treatment zone.
* Endoscopically visible abnormalities such as masses or nodules requiring endoscopic resection.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2015-01; Primary Completion 2016-12-29 (Actual); Study Completion 2017-10-04 (Actual)

PRIMARY OUTCOMES:
Presence of residual Barrett's Esophagus | 12 weeks
  Efficacy (% of) Barrett's epithelium fully converted to squamous epithelium upon cryoablation

SECONDARY OUTCOMES:
Incidence of adverse events | 12 weeks
  All adverse events will be reported
Patient Pain | post-procedure through 12 week follow-up
  Patient is asked to rate any pain in the treatment area or with swallowing
Device Performance | 12 weeks
  All device performance will be reported

CONTACTS AND LOCATIONS:
Overall Officials: Jacques Bergman, MD, PhD, Principal Investigator — Academic Medical Centre (Amsterdam)
Locations (2):
- Netherlands (2):
  - Academic Medical Center Amsterdam, Amsterdam
  - St. Antonius Hospital, Nieuwegein

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Friedland S, Triadafilopoulos G. A novel device for ablation of abnormal esophageal mucosa (with video). Gastrointest Endosc. 2011 Jul;74(1):182-8. doi: 10.1016/j.gie.2011.03.1119. Epub 2011 Apr 30. PMID 21531411
- [Derived] van Munster SN, Overwater A, Haidry R, Bisschops R, Bergman JJGHM, Weusten BLAM. Focal cryoballoon versus radiofrequency ablation of dysplastic Barrett's esophagus: impact on treatment response and postprocedural pain. Gastrointest Endosc. 2018 Nov;88(5):795-803.e2. doi: 10.1016/j.gie.2018.06.015. Epub 2018 Jun 19. PMID 29928869